CLINICAL TRIAL: NCT01189474
Title: Phase IV Multicentric Study, 140 Patients Suffering of Meibomian Glands Dysfunction.
Brief Title: Evaluation of Satisfaction Regarding Patient's Management of Ocular Surface Diseases
Acronym: ESPOIR Ext
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT2420-PIV-CE-02/10; N° RCB 2010-A00199-30 (Other: AFSSAPS)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Eyelid Diseases
Keywords: Meibomian Gland Dysfunction
MeSH Terms: conditions — Eyelid Diseases; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Blephasteam — Eye lid warming goggles

SUMMARY:
Multicentric study, open label, uncontrolled phase IV in 140 patients with meibomian glands dysfunction .

Its objective is to Collect information from patients and ophthalmologists specialized in ocular surface and eyelids to anticipate how Blephasteam ® can be optimized.

This study involves 2 visits, visit of Inclusion, J0, then end of study visit, D21.

Between the two visits patients will be treated with Blephasteam ® for 21 days (up to two uses per day) and complete a questionnaire every two days during the first week and then once a week the next two weeks.

ELIGIBILITY:
* Signed and dated informed consent.
* Male or female up to 4 years old.
* Known and treated symptomatic Meibomian Gland Diseases, and/or Dry Eye related to MGDs stable since at least a month.
* Without any active pathology requiring a change in ocular treatments within the last month before inclusion.
* Best corrected far visual acuity (VA) > 1/10

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul ADENIS, Professor, Principal Investigator — Hopital Dupuytren Limoges; Isabelle BADELLON, Doctor, Principal Investigator — Fondation Rothschild Paris; Vincent BORDERIE, Professor, Principal Investigator — CHNO des quinze-vingts; Tristan BOURCIER, Professor, Principal Investigator — CHU de Strasbourg; Jean Louis BOURGES, Doctor, Principal Investigator — Hotel Dieu Paris; Dominique BREMOND GIGNAC, Professor, Principal Investigator — Centre Hospitalier Universitaire, Amiens; Carole BURILLON, Professor, Principal Investigator — Hopital Edouard Heriot Lyon; Philippe CAZEMIND, Doctor, Principal Investigator — Clinique du cours Dillion; Hervé CHENAL, Doctor, Principal Investigator; Joseph COLIN, Professor, Principal Investigator — University Hospital, Bordeaux; Catherine CREUZOT GARCHER, Professor, Principal Investigator — Centre Hospitalier Universitaire Dijon; Stephan FAUQUIER, Doctor, Principal Investigator; Denis FLORES, Doctor, Principal Investigator; Philippe GAIN, Professor, Principal Investigator — CHU de Saint Etienne; Olivier Galatoire, Doctor, Principal Investigator — Fondation Rothschild Paris; Damien GATINEL, Doctor, Principal Investigator — Fondation Rothschild Paris; Jean Luc GEORGES, Professor, Principal Investigator — Central Hospital, Nancy, France; Thanh HOANG XUAN, Professor, Principal Investigator; Philippe IMBERT, Doctor, Principal Investigator — Polyclinique du Parc; Marc LABETOULLE, Professor, Principal Investigator — CH de Bicetre; Karim LAOUAR, Doctor, Principal Investigator — Centre Hospitalier de Nimes; Sylvie MAES CASTELLARIN, Doctor, Principal Investigator — Hopital de Tarbes; Sylvie MAINGUY, Doctor, Principal Investigator; Claire MEURIOT TUIL, Doctor, Principal Investigator; Solange MILAZZO, Professor, Principal Investigator — Centre Hospitalier Universitaire, Amiens; Bruno MORTEMOUSQUE, Doctor, Principal Investigator — University Hospital, Bordeaux; Pierre Jean PISELLA, Professor, Principal Investigator — CHU de Tours; Pierre Yves ROBERT, Professor, Principal Investigator — University Hospital, Limoges; Stephane RONCIN, Doctor, Principal Investigator — Polyclinique Saint Laurent; Jean François ROULAND, Professor, Principal Investigator — CHU de Lille; Pierre LABALETTE, Professor, Principal Investigator — CHU de Lille; Frank ROUX, Doctor, Principal Investigator — HIA Laveran; Claude SPEEG, ¨Professor, Principal Investigator — CHU de Strasbourg; Michel TAZARTES, Doctor, Principal Investigator; Yves UTEZA, Doctor, Principal Investigator; Hatem ZEGHIDI, Doctor, Principal Investigator; Benoit BRIAT, Doctor, Principal Investigator
Locations (29):
- France (29):
  - CHU d'Amiens, Amiens
  - Hopital Pellegrin, Bordeaux
  - CHU de Dijon, Dijon
  - 76 Allée des Pins Tranquilles, Hossegord
  - CHU de BicÃªtre, Le Kremlin BicÃªtre
  - Hopital Claude Huriez, Lille
  - Hopital Dupuytren, Limoges
  - Hopital Edouard Heriot, Lyon
  - 433 bis rue Paradis, Marseille
  - Hopital d'instruction des armées LAVERAN, Marseille
  - 67 chemin du Fescau, Montferrier-sur-Lez
  - 60 place Jacques Mirouze, Montpellier
  - 3 cours Leopold, Nancy
  - Hopital Max Fourestier, Nanterre
  - 4 avenue Baquis, Nice
  - Centre Hospitalier de Nimes, Nîmes
  - 22 rue Beaujon, Paris
  - Hotel Dieu, Paris
  - C.H.N.O des XV-XX, Paris
  - 142 Boulevard de Montparnasse, Paris
  - Fondation Rothschild, Paris
  - 26 rue du Moulin des justices, Puilboreau
  - Polyclinique Saint Laurent, Rennes
  - CHU de Saint Etienne, Saint-Etienne
  - CHU Hospices Civils, Strasbourg
  - Hôpital de Tarbes, Tarbes
  - Clinique du Cours Dillion, Toulouse
  - CHU Bretonneau, Tours
  - Hopital Brabois Adulte, Vandœuvre-lès-Nancy